CLINICAL TRIAL: NCT00064298
Title: A Phase II Randomized Placebo Controlled, Double Blinded Trial To Evaluate The Effects Of Fruit And Vegetable Extracts On Intermediate Biomarkers In Head And Neck Cancer Patients
Brief Title: Fruit and Vegetable Extracts in Treating Patients With Stage I-IV, Stage IVA/IVB Head and Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: REBAWFU-60A02; U10CA081851 (NIH)
Record Dates: First submitted 2003-07-08; First posted 2003-07-09 (Estimated); Results first posted 2017-07-24 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Head and Neck Cancer
Keywords: stage I squamous cell carcinoma of the hypopharynx; stage I squamous cell carcinoma of the larynx; stage I squamous cell carcinoma of the lip and oral cavity; stage I squamous cell carcinoma of the oropharynx; stage II squamous cell carcinoma of the hypopharynx; stage II squamous cell carcinoma of the larynx; stage II squamous cell carcinoma of the lip and oral cavity; stage II squamous cell carcinoma of the oropharynx; stage III squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the larynx; stage III squamous cell carcinoma of the lip and oral cavity; stage III squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the oropharynx
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Fruit

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I - JuicePlus (Experimental): Patients receive oral fruit and vegetable extracts twice daily.
  Interventions: Dietary Supplement: fruit and vegetable extracts
- Arm II - Control (Placebo Comparator): Patients receive oral placebo twice daily.
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: fruit and vegetable extracts — Given orally
  Arms: Arm I - JuicePlus
Dietary Supplement: placebo — Given orally
  Arms: Arm II - Control

SUMMARY:
RATIONALE: Chemoprevention therapy is the use of certain substances to try to prevent the development or recurrence of cancer. Fruit and vegetable extracts may be effective in preventing the recurrence or further development of head and neck cancer.

PURPOSE: This randomized phase II trial is studying how well fruit and vegetable extracts work in preventing the recurrence of stage I, stage II, stage III, stage IVA, or stage IVB head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the disease-free survival of patients with stage I-IV (including stage IVA and IVB) head and neck cancer treated with fruit and vegetable extracts vs placebo.
* Compare the effect of these extracts on biomarkers (p27 expression, cell proliferation of Ki-67, DNA damage, and T-cell function) in these patients.
* Correlate changes in biomarkers with other factors (e.g., site and stage of the original tumors, tobacco/alcohol use, or depression) in patients treated with these extracts.
* Compare serum carotenoids and antioxidant levels (vitamins A, C, and E) at baseline and posttreatment in patients treated with these extracts.

OUTLINE: This is a randomized, placebo-controlled, double-blind study. Patients are stratified according to tobacco use (yes vs no), alcohol consumption (yes vs no), and tumor stage at diagnosis (I vs II vs III vs IVA vs IVB). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral fruit and vegetable extracts twice daily.
* Arm II: Patients receive oral placebo twice daily. Treatment in both arms continues for 12 weeks in the absence of disease progression or unacceptable toxicity.

Patients are followed annually for 5 years.

PROJECTED ACCRUAL: A total of 200 patients (100 per treatment arm) will be accrued for this study within 18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Curatively treated stage I-IV (including stage IVA and IVB) squamous cell carcinoma of the upper aerodigestive tract of 1 of the following primary sites:

  * Oral cavity
  * Oropharynx
  * Hypopharynx
  * Larynx
* Disease-free for at least 6 months and no more than 3 years after completion of surgery, radiotherapy, and/or chemotherapy
* No synchronous tumors

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Karnofsky 70-100% OR
* Zubrod 0-1

Life expectancy

* At least 6 months

Hematopoietic

* Hemoglobin ≥ 10 g/dL
* WBC ≥ 3,000/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* Bilirubin ≤ 1.5 mg/dL
* SGOT ≤ 40 U/L
* SGPT ≤ 56 U/L

Renal

* Creatinine ≤ 1.5 mg/dL

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other malignancy within the past 5 years except curatively treated head and neck squamous cell carcinoma, nonmelanoma skin cancer, or carcinoma in situ of the cervix
* No other serious medical or psychiatric illness that would preclude giving informed consent
* No nausea ≥ grade 2

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* See Disease Characteristics
* More than 6 months and less than 3 years since prior chemotherapy
* No concurrent chemotherapy
* No other concurrent chemopreventive agents

Endocrine therapy

* More than 6 months and less than 3 years since prior hormonal therapy

Radiotherapy

* See Disease Characteristics
* More than 6 months and less than 3 years since prior radiotherapy
* No concurrent radiotherapy

Surgery

* See Disease Characteristics
* More than 6 months and less than 3 years since prior surgery
* No concurrent surgery

Other

* More than 6 months and less than 3 years since prior investigational agents
* More than 2 months since prior high-dose vitamins (i.e., 10 times the recommended daily allowance [8,000-10,000 IU of vitamin A, 600 mg of vitamin C, or 80-100 IU of vitamin E])

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2004-01-01 (Actual); Primary Completion 2008-10-01 (Actual); Study Completion 2009-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven A. Akman, MD, Study Chair — Wake Forest University Health Sciences
Locations (28):
- United States (28):
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - Redwood Regional Medical Group, Santa Rosa, California
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - MBCCOP - Howard University Cancer Center, Washington D.C., District of Columbia
  - University of Miami Sylvester Comprehensive Cancer Center - Miami, Miami, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - MBCCOP - JHS Hospital of Cook County, Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Feist-Weiller Cancer Center at Louisiana State University Health Sciences, Shreveport, Louisiana
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - CCOP - Beaumont, Royal Oak, Michigan
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - Alamance Cancer Center at Alamance Regional Medical Center, Burlington, North Carolina
  - Hugh Chatham Memorial Hospital, Elkin, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Goldsboro, North Carolina
  - Leo W. Jenkins Cancer Center at ECU Medical School, Greenville, North Carolina
  - High Point Regional Hospital, High Point, North Carolina
  - Caldwell Memorial Hospital, Lenoir, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Danville Regional Medical Center, Danville, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Datta M, Shaw EG, Lesser GJ, Case LD, Vitolins MZ, Schneider C, Frizzell B, Sullivan C, Lively M, Franzmann E, Hu JJ. A Randomized Double-Blind Placebo-Controlled Trial of Fruit and Vegetable Concentrates on Intermediate Biomarkers in Head and Neck Cancer. Integr Cancer Ther. 2018 Mar;17(1):115-123. doi: 10.1177/1534735416684947. Epub 2017 Jan 19. PMID 28102098

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants are recruited from NCI CCOP sites.
Period: Overall Study
Arm/Group | Arm I - JuicePlus | Arm II - Control
Started | 72 | 62
Completed | 66 | 57
Not Completed | 6 | 5
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Lost to Follow-up | 2 | 2
Not completed — Death | 0 | 1
Not completed — Disease Progression | 2 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I - JuicePlus | Arm II - Control | Total
Number analyzed (Participants) | 72 | 62 | 134
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 51 | 46 | 97
  >=65 years | 21 | 16 | 37
Age, Continuous [Median (Full Range); unit: years] | 58 [30 to 82] | 59 [41 to 82] | 58 [30 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 21
  Male | 61 | 52 | 113
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 2 | 9
  Not Hispanic or Latino | 64 | 60 | 124
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 7 | 11
  White | 64 | 55 | 119
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 0 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 72 | 62 | 134

OUTCOME MEASURES:

1. Primary Outcome: Expression of p27 Cell Cycle Regulatory Protein at Baseline and Week 12
Description: Expression of p27 cell cycle regulatory protein at baseline and week 12. p27 is measured continuously. Lower values are worse.
Time Frame: baseline and 12 weeks
Population: All randomized participants. Not all participants had p27 or Ki67 determined, so the sample sizes for the two outcomes differ from the total sample size.
Measure: Mean (Standard Error); unit: percentage of cells
Arm/Group | Arm I - JuicePlus | Arm II - Control
Number analyzed (Participants) | 72 | 62
percentage of cells
  Baseline: number analyzed (Participants) | 54 | 45
  Baseline | 18.6 (1.52) | 15.1 (1.42)
  12 weeks: number analyzed (Participants) | 57 | 62
  12 weeks | 17.0 (1.39) | 14.5 (1.57)

2. Secondary Outcome: Cell Proliferation (Ki-67) at Baseline and Week 12
Description: Cell proliferation (Ki-67) at baseline and week 12. Ki67 is a cell proliferation associated nuclear protein. It is measured continuously. Higher values are worse.
Time Frame: baseline and 12 weeks
Population: All participants randomized. Not all participants had p27 or Ki67 data so the sample sizes for the primary and secondary analyses differ from the overall sample size.
Measure: Mean (Standard Error); unit: percentage of cells
Arm/Group | Arm I - JuicePlus | Arm II - Control
Number analyzed (Participants) | 72 | 62
percentage of cells
  Baseline: number analyzed (Participants) | 45 | 42
  Baseline | 26.8 (1.20) | 26.2 (1.28)
  12 Weeks: number analyzed (Participants) | 47 | 40
  12 Weeks | 27.1 (1.43) | 27.0 (1.55)

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Sample size is number of participants with follow-up toxicity data recorded.
Arm/Group | Arm I - JuicePlus | Arm II - Control
Serious Adverse Events (participants affected / at risk) | 2/68 | 2/59
Other Adverse Events (participants affected / at risk) | 21/68 | 16/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I - JuicePlus (N=68) | Arm II - Control (N=59)
Dehydration (Gastrointestinal disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 2 (2) | 0 (0)
Ataxia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Mood Change (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 4.4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I - JuicePlus (N=68) | Arm II - Control (N=59)
Diarrhea (Gastrointestinal disorders) | 4 (5) | 4 (5)
Dysphagia (Musculoskeletal and connective tissue disorders) | 4 (5) | 0 (0)
Fatigue (Metabolism and nutrition disorders) | 3 (7) | 2 (7)
Gas (Gastrointestinal disorders) | 0 (0) | 3 (4)
Heartburn (Gastrointestinal disorders) | 7 (7) | 6 (12)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (3)
Pain (General disorders) | 3 (3) | 3 (3)
SOB (General disorders) | 4 (4) | 0 (0)
Taste Alteration (General disorders) | 3 (11) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes